CLINICAL TRIAL: NCT01793571
Title: A Pilot Study on the Effectiveness of the Echoguided Transversus Abdominis Plane Block During Inguinal Hernia Repair Surgery
Brief Title: Pilot Study on the Effectiveness of a TAP-block for Inguinal Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dijklander Ziekenhuis (Other)
Responsible Party: Principal Investigator, Peter Dijkhuizen, MPA Anesthesiology, Dijklander Ziekenhuis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL40460.094.12
Record Dates: First submitted 2013-01-17; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Hernia Inguinal
Keywords: Abdominal Muscles/Ultrasonography; Adult; Ambulatory Surgical Procedures; Anesthetics, Local/Administration & Dosage; Levobupivacaine/Administration & Dosage; Levobupivacaine/Analogs & Derivatives; Hernia, Inguinal/Surgery; Humans; Nerve Block/Methods; Pain Measurement/Methods; Pain, Postoperative/Prevention & Control; Ultrasonography, Interventional
MeSH Terms: conditions — Hernia, Inguinal; Hernia; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP block (Experimental): 20 ml Levobupivacaine 0,5%
  Interventions: Procedure: TAP block
- Local wound infiltration (Active Comparator): 20 ml levobupivacaine 0,5%
  Interventions: Procedure: TAP block

INTERVENTIONS:
Procedure: TAP block — 2 groups, group A a TAP block with 20 ml of Levobupivacaine 0,5% and subcutaneous wound infiltration with 20 ml sodium chloride (to blind patient and physician) and group B, TAP block with 20 ml sodium chloride and subcutaneous wound infiltration with 20 ml Levobupivacaine 0,5% (to blind patient and physician)

SUMMARY:
An prospective double blinded randomised trial,whether the use of an perioperative echoguided unilateral TAP block has an superior effect on postoperative pain after open hernia inguinal repair compared to wound infiltration with a long acting local anesthetic.

DETAILED DESCRIPTION:
Hernia inguinal repair is the most common operation performed by general surgeons in the Netherlands. On of the most common complications after hernia repair is postoperative and chronic pain. Postoperative pain is an expected but undesirable effect after an operation, which can result in an prolonged hospital stay or longer time to return to full normal daily activities. There are indications that an insufficient treatment of postoperative pain is a risk factor for persistent or chronic pain after open inguinal hernia repair. Chronic pain is not uncommon after hernia repair, with an incidence of 11%.

The objective of this study is to determine, whether the use of an perioperative echo guided unilateral TAP block has an superior effect on postoperative pain after open hernia inguinal repair compared to wound infiltration with a long acting local anesthetic. There will be no further analysis in this study regarding the incidence of open hernia inguinal repair and chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 year, competent, elective surgical treatment, Body Mass Index (BMI) between 20-35.

Exclusion Criteria:

* fever, a coagulation disorder, patients with kidney and liverfaillure, an infection at the place where the puncture place, preoperative use of narcotic and nonsteroidal antiinflammatory drugs.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Primary objective is to analyse, differences in pain scores between the 2 groups until 48 hours after the operation | 48 hours

SECONDARY OUTCOMES:
time to to first use of intravenous morfine | 48 hours
the total amount of titrated postoperative morfine | 48 hours
use of tramadol at home | 48 hours
patient satisfaction | 48 hours
the incidence of nausea and vomiting | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jens P Hering, Anesthesiologist, Principal Investigator — Dijklander Ziekenhuis
Locations (1):
- Westfriesgasthuis, Hoorn, North Holland, Netherlands